CLINICAL TRIAL: NCT00549536
Title: The Effect of Oral Calcium Supplementation on Insulin Sensitivity, Intracellular Cationic Concentrations and the Transmembrane Sodium/Hydrogen Exchanger Activity in Subjects With Type 2 Diabetes and Hypertension
Brief Title: The Effect of Calcium Supplementation on Insulin Resistance and 24h Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Hellenic Society of Hypertension (Other)
Responsible Party: Lasaridis Anastasios, 1st Department of medicine AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A3242
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension; Diabetes; Insulin Resistance
Keywords: calcium supplementation; intracellular ions; sodium/hydrogen exchange activity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Insulin Resistance | interventions — Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention)
  Interventions: Dietary Supplement: tablets each containing of 1000mg elemental calcium (Mega-Calcium Sandoz)
- 1 (Active Comparator): Patients on calcium supplementation
  Interventions: Dietary Supplement: tablets each containing of 1000mg elemental calcium (Mega-Calcium Sandoz)

INTERVENTIONS:
Dietary Supplement: tablets each containing of 1000mg elemental calcium (Mega-Calcium Sandoz) — 1500 mg of elemental calcium per day.
  Other Names: Mega-Calcium Sandoz

SUMMARY:
Increased levels of intracellular calcium are thought to diminish maximal cellular response to insulin and induce insulin resistance. Also, both hypertension and diabetes are thought to be conditions of altered intracellular ionic state. The aim of the present study is to investigate the possible effect of oral calcium supplementation on intracellular ions, insulin sensitivity, 24-h blood pressure and sodium/hydrogen exchanger activity in patients with type 2 diabetes and essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension, diabetes and the metabolic syndrome (according to the definition of the National Cholesterol Education Program, Adult Panel III (NCEP, ATP III).
* Signed the concent form

Exclusion Criteria:

* Secondary Hypertension
* Stage II or III hypertension
* History of renal disease
* Sleep apnea
* Acute or chronic inflammation
* History of coronary artery disease
* Heart failure stage III or IV according to the New York Heart Association
* Active liver disease
* History of malignancy
* Parathyroidism
* History of kidney stones
* Calcium supplement ingestion
* Drugs that alter insulin resistance
* Treatment with insulin
* Alcohol abuse or other conditions with poor prognosis
* Treatment with non-inflammatory steroid agents, corticosteroids, or any other treatment that affects blood pressure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the difference in 24h blood pressure measurement and insulin sensitivity between the treatment and the control group. | baseline and after 8 weeks of follow up

SECONDARY OUTCOMES:
To evaluate differences in intracellular calcium, magnesium, sodium and potassium concentrations at the end of the follow up period between the calcium supplementation group and the control group. | baseline and after 8 weeks of follow up
To evaluate differences in the transmembrane sodium/hydrogen exchanger activity between the active treatment and the control group. | baseline and after 8 weeks of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios N. Lasaridis, MD, PhD, Principal Investigator — 1st Department of Internal Medicine, AHEPA University Hospital, Aristotle University of Thessaloniki, Greece; Maria I. Pikilidou, MD, MSc, Study Director — 1st Department of Internal Medicine, AHEPA University Hospital, Aristotle University of Thessaloniki, Greece
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece